CLINICAL TRIAL: NCT05194566
Title: Neurostimulation for the Treatment of Post-Stroke Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro Device S.A (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-21-01577
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-07

CONDITIONS: Post-stroke Aphasia
Keywords: speech therapy; brain stimulation; communication; language
MeSH Terms: conditions — Communication Disorders; Communication; Language | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The study will employ a between-subject randomized sham-controlled design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, investigator and outcomes assessor are all blinded. Designated research team members will be unblinded in order to manage computerized procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Real tACS (Active Comparator): tACS 75Hz intervention combined with language tasks and breathing exercises. The device will operate in tACS research active stimulation mode.
  Interventions: Device: tACS
- Sham tACS (Sham Comparator): tACS sham intervention combined with language tasks and breathing exercises. The device will operate in tACS sham simulation research mode.
  Interventions: Device: tACS

INTERVENTIONS:
Device: tACS — Neurostimulation will be done using the Neuro Device tCS (Neuro Device tCS), which is a certified transcranial electrical stimulator. The device consists of a stimulator with a touch screen, two electrodes and a soft, flexible cap to ensure stability of the electrodes on the head.
  Other Names: transcranial alternating current stimulation

SUMMARY:
The aim of the trial is to determine whether 75Hz transcranial alternating current stimulation (tACS) synchronized with therapeutic linguistic tasks is an effective form of therapy for post-stroke aphasia.

DETAILED DESCRIPTION:
There are about 15 million strokes worldwide each year. Of this group, about 30% suffer from aphasia. Aphasia is a speech-language disorder associated with exceptional difficulty performing daily communication activities. If no improvement is observed within the first months after the stroke, a complete recovery is unlikely, and the therapy can last for years.

Up to date, speech and language therapy is a standard of care for post-stroke aphasia, however the process is long and demanding.

In the past, several clinical trials aimed to verify the efficacy of language training paired with transcranial direct current stimulation (tDCS), however recent meta-analysis indicates only possible effectiveness (Level C evidence) of anodal tDCS in chronic post-stroke aphasia.

To boost the effects of aphasia rehabilitation, effective brain stimulation protocol still needs to be developed.

Transcranial alternating current stimulation (tACS) can be an interesting alternative to tDCS, as it is able to influence cortical excitability and activity.

Stimulation within high gamma oscillations (60-500Hz) might allow for better speech-language processing, as this band is considered to be the cognitive index of linguistic processes. Moreover, a short period of 75Hz tACS over the motor cortex suggested the positive impact of high-gamma tACS on brain plasticity.

The aim of this RCT is to determine whether 75Hz transcranial alternating current stimulation (tACS) paired with therapeutic linguistic tasks is an effective form of therapy for post-stroke aphasia, measured as an ability to name trained items at 12 weeks follow-up.

ELIGIBILITY:
Individuals with aphasia (assessed using the Boston Diagnostic Aphasia Examination) who perform the Naming Task in the range of 10%-60% accuracy will be included in the study. The overall baseline score in the Naming Task will be estimated from the two baseline measurements.

Inclusion Criteria:

* diagnosis of aphasia: Broca's or mixed (based on the assessment of a Speech Language Pathologist).
* presence of a focus of injury in the left hemisphere (within one hemisphere only) as a result of the first ischemic or hemorrhagic stroke (based on CT/MRI examination);
* chronic stage of the disease - time since the stroke occurred over 6 months.
* ability to achieve an accuracy in the Naming Task of 10-60%.
* 18-80 years
* right-handedness before the stroke.
* ability to give informed written consent.
* fluency in English.

Exclusion Criteria:

* severe cognitive, auditory or visual impairment that would preclude cognitive and language testing - inability to follow a two-step command.
* presence of metal implants in the skull.
* presence of major untreated or unstable psychiatric disease.
* history of epilepsy or seizures.
* ongoing medication that increases the risk of epileptic seizures.
* presence in the body of cardiac stimulators or pacemaker.
* history of speech, language, hearing, or intellectual disability during childhood.
* pregnancy (based on declarations)

Exclusion criteria during the trial:

* high intolerance to stimulation.
* occurrence of an epileptic seizure.
* other previously absent neurological or mental symptoms

Withdrawal criteria:

* high intolerance to stimulation (participants experience severe discomfort during stimulation);
* occurrence of an epileptic seizure;
* other previously absent neurological, physical or mental symptoms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage score in the Naming Task (trained words) | at 12 weeks
  The Baseline Naming Task consists of 344 images representing nouns and the images will be presented on the computer screen. The task is to name the presented noun by producing the name of the item out loud. The answer is scored on a three-point scale (1 - not able to name correctly, 2 - named with phonological or semantic paraphasia, 3 - correct). Items marked with a score of 3 are considered accurate. From the baseline assessment, a random list of 50 incorrectly named words will be trained in therapy. Minimum score is 0% (inability to name any objects) and maximum score is 100% (accuracy in naming all presented objects), where a higher score indicates a better health outcome

SECONDARY OUTCOMES:
Naming Task (untrained words) | at 12 weeks
  Generalization - percentage score in the Naming Task (untrained words). The answer is scored on a three-stage scale (1 - not able to name correctly, 2 - named with phonological or semantic paraphasia, 3 - correct). Every Naming Task session will be recorded, so the independent SLP (speech-language pathologist) will again assess response accuracy. In case of inconsistency of scores, third independent SLP will decide.
Naming reaction time (within baseline naming task) | at Baseline
  Amount of time elapsed between the presentation of the stimuli to the first attempt of the patient's response. Measured by clinician recording of time elapsed before response attempted for each stimuli presented. Average overall response time will at baseline will be recorded.
Naming reaction time (within baseline naming task) | at 12-week follow-up
  Amount of time elapsed between the presentation of the stimuli to the first attempt of the patient's response. Measured by clinician recording of time elapsed before response attempted for each stimuli presented. Average overall response time at 12-week follow-up will be recorded.
Number of correct answers without supporting cues | 2 weeks
  Number of correct answers on the fifth level (no cueing) during the therapy task. Greater number of correct responses indicates better response to treatment.
Accuracy of naming during the therapy session | 2 weeks
  Number of correct responses to presented stimuli. Greater number of correct responses indicates better response to treatment.
Percentage Score in Naming Task (untrained words) | at Baseline
  Percentage score calculated for words not trained in therapy task to assess generalization. Patients are presented with 25 words not trained during therapy sessions. Each answer is scored on a three-point scale (1 - not able to name correctly, 2 - named with phonological or semantic paraphasia, 3 - correct). Items receiving a score of 3 are marked as correct, with a maximum total number of correct items being 25. Minimum score is 0% (0/25- inability to name any objects) and maximum score is 100% (25/25- accuracy in naming all presented objects), where higher score indicates better response to treatment.
Percentage Score in Naming Task (untrained words) | at the end of the last therapy session at the end of week 4
  Percentage score calculated for words not trained in therapy task to assess generalization. Patients are presented with 25 words not trained during therapy sessions. Each answer is scored on a three-point scale (1 - not able to name correctly, 2 - named with phonological or semantic paraphasia, 3 - correct). Items receiving a score of 3 are marked as correct, with a maximum total number of correct items being 25. Minimum score is 0% (0/25- inability to name any objects) and maximum score is 100% (25/25- accuracy in naming all presented objects), where higher score indicates better response to treatment.
Percentage Score in Naming Task (untrained words) | at 6-week follow-up
  Percentage score calculated for words not trained in therapy task to assess generalization. Patients are presented with 25 words not trained during therapy sessions. Each answer is scored on a three-point scale (1 - not able to name correctly, 2 - named with phonological or semantic paraphasia, 3 - correct). Items receiving a score of 3 are marked as correct, with a maximum total number of correct items being 25. Minimum score is 0% (0/25- inability to name any objects) and maximum score is 100% (25/25- accuracy in naming all presented objects), where higher score indicates better response to treatment.
Percentage Score in Naming Task (untrained words) | at 12-week follow-up
  Percentage score calculated for words not trained in therapy task to assess generalization. Patients are presented with 25 words not trained during therapy sessions. Each answer is scored on a three-point scale (1 - not able to name correctly, 2 - named with phonological or semantic paraphasia, 3 - correct). Items receiving a score of 3 are marked as correct, with a maximum total number of correct items being 25. Minimum score is 0% (0/25- inability to name any objects) and maximum score is 100% (25/25- accuracy in naming all presented objects), where higher score indicates better response to treatment.
Communication Effectiveness Index (CETI) | at Baseline
  The participants primary communication partner rates the participants' ability to perform in sixteen communication situations on a visual analog scale with the lowest value (a score of 0) as "not at all able" and the greatest value (a score of 10) as "as able to as before", where higher scores indicate better health outcomes.
Communication Effectiveness Index (CETI) | at the end of the last therapy session at the end of week 4
  The participants primary communication partner rates the participants' ability to perform in sixteen communication situations on a visual analog scale with the lowest value (a score of 0) as "not at all able" and the greatest value (a score of 10) as "as able to as before", where higher scores indicate better health outcomes.
Communication Effectiveness Index (CETI) | at 6-week follow-up
  The participants primary communication partner rates the participants' ability to perform in sixteen communication situations on a visual analog scale with the lowest value (a score of 0) as "not at all able" and the greatest value (a score of 10) as "as able to as before", where higher scores indicate better health outcomes.
Communication Effectiveness Index (CETI) | at 12-week follow-up
  The participants primary communication partner rates the participants' ability to perform in sixteen communication situations on a visual analog scale with the lowest value (a score of 0) as "not at all able" and the greatest value (a score of 10) as "as able to as before", where higher scores indicate better health outcomes.
Boston Diagnostic Aphasia Examination (BDAE) | at Baseline
  Oral Expression Subtest - the speech language pathologist assesses the patient with the oral expression portion of the BDAE. Areas assessed include automatic sequences, repetition of words and sentences, responsive and confrontational naming, and screening of letters and numbers. Each item receives a point for correctness with a maximal score of 48
Boston Diagnostic Aphasia Examination (BDAE) | at 12-week follow-up
  Oral Expression Subtest - the speech language pathologist assesses the patient with the oral expression portion of the BDAE. Areas assessed include automatic sequences, repetition of words and sentences, responsive and confrontational naming, and screening of letters and numbers. Each item receives a point for correctness with a maximal score of 48
Accuracy of masking measurement: Patient and Researcher | end of treatment (at 12 weeks)
  The opinion of the patient and of the researcher on receiving the placebo vs. active stimulation. The patient and researcher provide their guess/opinion as to whether the stimulation received during treatment was active or sham. It will be taken after the end of the last treatment session.
Visual Analog Scale (VAS) | 2 weeks
  Stimulation tolerance/side effects are measured using a visual analog scale with seven components (headache, fatigue, sleepiness, dizziness, pain on scalp, tingling on scalp, burning sensation on scalp, and itching on scalp). Ratings will be taken before and after each session. Full scale 0-10 per component. Higher score indicates a higher degree of each side effect.
Stroke and Aphasia Quality of Life Scale (SAQOL-39) Score | at Baseline
  Assesses the ability to complete daily tasks pertaining to self-care, communication, interaction with others, and physical mobility. The SAQOL includes 17 questions, where questions are rated on a 1-5 scale with a score of 1 indicating greater disability and 5 indicating none. Total score ranges from 17-85. Scores are averaged across three domains (physical, communication, and psychosocial), with lower scores indicating lesser ability (lower quality of life) and higher scores indicating great ability or independence (greater quality of life)
Stroke and Aphasia Quality of Life Scale (SAQOL-39) Score | at the end of the last therapy session at the end of week 4
  Assesses the ability to complete daily tasks pertaining to self-care, communication, interaction with others, and physical mobility. The SAQOL includes 17 questions, where questions are rated on a 1-5 scale with a score of 1 indicating greater disability and 5 indicating none. Total score ranges from 17-85. Scores are averaged across three domains (physical, communication, and psychosocial), with lower scores indicating lesser ability (lower quality of life) and higher scores indicating great ability or independence (greater quality of life)
Stroke and Aphasia Quality of Life Scale (SAQOL-39) Score | at 6-week follow-up
  Assesses the ability to complete daily tasks pertaining to self-care, communication, interaction with others, and physical mobility. The SAQOL includes 17 questions, where questions are rated on a 1-5 scale with a score of 1 indicating greater disability and 5 indicating none. Total score ranges from 17-85. Scores are averaged across three domains (physical, communication, and psychosocial), with lower scores indicating lesser ability (lower quality of life) and higher scores indicating great ability or independence (greater quality of life)
Stroke and Aphasia Quality of Life Scale (SAQOL-39) Score | at 12-week follow-up
  Assesses the ability to complete daily tasks pertaining to self-care, communication, interaction with others, and physical mobility. The SAQOL includes 17 questions, where questions are rated on a 1-5 scale with a score of 1 indicating greater disability and 5 indicating none. Total score ranges from 17-85. Scores are averaged across three domains (physical, communication, and psychosocial), with lower scores indicating lesser ability (lower quality of life) and higher scores indicating great ability or independence (greater quality of life)
General Health Questionnaire (GHQ-12) | at Baseline
  Identifies minor psychiatric disorders in the general population and within community or non-psychiatric clinical settings such as primary care or general medical out-patients. GHQ-12 is a 12-items scaled version that assesses somatic symptoms, anxiety, and insomnia, social dysfunction, and severe depression. A total score ranges from 0 to 36, with higher scores indicating worse conditions
General Health Questionnaire (GHQ-12) | at the end of the last therapy session at the end of week 4
  Identifies minor psychiatric disorders in the general population and within community or non-psychiatric clinical settings such as primary care or general medical out-patients. GHQ-12 is a 12-items scaled version that assesses somatic symptoms, anxiety, and insomnia, social dysfunction, and severe depression. A total score ranges from 0 to 36, with higher scores indicating worse conditions
General Health Questionnaire (GHQ-12) | at 6-week follow-up
  Identifies minor psychiatric disorders in the general population and within community or non-psychiatric clinical settings such as primary care or general medical out-patients. GHQ-12 is a 12-items scaled version that assesses somatic symptoms, anxiety, and insomnia, social dysfunction, and severe depression. A total score ranges from 0 to 36, with higher scores indicating worse conditions
General Health Questionnaire (GHQ-12) | at 12-week follow-up
  Identifies minor psychiatric disorders in the general population and within community or non-psychiatric clinical settings such as primary care or general medical out-patients. GHQ-12 is a 12-items scaled version that assesses somatic symptoms, anxiety, and insomnia, social dysfunction, and severe depression. A total score ranges from 0 to 36, with higher scores indicating worse conditions
Brief Resilience Scale (BRS) | at Baseline
  Assesses the perceived ability to bounce back or recover from stress. The possible score range on the BRS is from 1 (low resilience) to 5 (high resilience). Higher scores indicate better health outcomes.
Brief Resilience Scale (BRS) | at the end of the last therapy session at the end of week 4
  Assesses the perceived ability to bounce back or recover from stress. The possible score range on the BRS is from 1 (low resilience) to 5 (high resilience). Higher scores indicate better health outcomes.
Brief Resilience Scale (BRS) | at 6-week follow-up
  Assesses the perceived ability to bounce back or recover from stress. The possible score range on the BRS is from 1 (low resilience) to 5 (high resilience). Higher scores indicate better health outcomes.
Brief Resilience Scale (BRS) | at 12-week follow-up
  Assesses the perceived ability to bounce back or recover from stress. The possible score range on the BRS is from 1 (low resilience) to 5 (high resilience). Higher scores indicate better health outcomes.
BDNF genotype | at Baseline
  Saliva samples will be collected to test for typical vs. atypical brain plasticity biomarkers, as BDNF genotype may interfere with results of therapy paired with transcranial electrical stimulation. Research suggests that individuals with an atypical BDNF genotype are less receptive to the beneficial effects of speech-language therapy paired with anodal transcranial direct current stimulation, compared to individuals with typical BDNF genotype

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Escalon, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Think & Speak Lab at Shirley Ryan AbilityLab, Chicago, Illinois
  - Abilities Research Center at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No
Not applicable to study aims

REFERENCES:
- [Background] Fridriksson J, Elm J, Stark BC, Basilakos A, Rorden C, Sen S, George MS, Gottfried M, Bonilha L. BDNF genotype and tDCS interaction in aphasia treatment. Brain Stimul. 2018 Nov-Dec;11(6):1276-1281. doi: 10.1016/j.brs.2018.08.009. Epub 2018 Aug 18. PMID 30150003